CLINICAL TRIAL: NCT05217706
Title: Low-Dose Intravenous Ketamine for Adolescents With Depression and Suicidal Ideation in the Emergency Department: A Randomized Placebo-Controlled Trial
Brief Title: Low-Dose Intravenous Ketamine for Adolescents With Depression and Suicidal Ideation in the Emergency Department
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rady Children's Hospital, San Diego (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Tanya Vayngortin, Assistant Clinical Professor, Rady Children's Hospital, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 800170
Record Dates: First submitted 2021-12-15; First posted 2022-02-01 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Depression; Suicidal Ideation
Keywords: emergency department; adolescent; ketamine
MeSH Terms: conditions — Depression; Suicidal Ideation; Emergencies | interventions — Ketamine; Saline Solution

STUDY DESIGN:
Intervention Model Description: double-blinded randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The enroller, treating provider, and patient are masked. Only the pharmacist will be un-masked, as they are preparing the medication or placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): This group will be given ketamine 0.2mg/kg
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator): This group will be given normal saline in matched syringe
  Interventions: Drug: normal Saline

INTERVENTIONS:
Drug: Ketamine — The treatment group will receive Ketamine 0.2mg/kg IV once
  Arms: Treatment
Drug: normal Saline — The placebo group will receive normal saline IV in a matched syringe
  Arms: Placebo

SUMMARY:
The goal of this study is to test whether a single low-dose of IV ketamine given in the emergency department to adolescents with treatment-resistant depression and suicidal ideation can reduce depression symptoms and suicidal thoughts compared to placebo. Participants will complete depression scales at baseline, and 1 hour, 3 hours, 1 day, 3 days, and 7 days after receiving the treatment.

DETAILED DESCRIPTION:
This study will be a double-blinded, randomized, placebo-controlled trial. Study investigators and trained research assistants (RAs) will identify eligible participants from the electronic ED tracking board based on inclusion criteria, and will confirm eligibility with the treating physician. After a patient has been evaluated by nursing, physician, and social worker and has been determined to require inpatient psychiatric admission, the patient and parent/guardian will be approached for the study. A parent/guardian must be available in person or by phone to provide consent, and the adolescent will provide assent. The RA or investigator will collect demographic data and psychiatric history from the electronic medical record to verify eligibility criteria, and will confirm with the treating physician that the patient can participate in the study. The RA or investigator will provide the patient self-administered scales, including the Suicidal Ideation Questionnaire and the Beck Depression, Anxiety, and Self-Concept Scales.

After the patient has assented and parent/guardian has consented to participation in the study, a study physician will initiate the electronic study order set. The Investigational Drug Service Pharmacy at RCHSD will dispense either ketamine 0.2 mg/kg (minimum 10 mg, maximum 20 mg) or normal saline in the same volume in identically-appearing syringe, based upon a pre-determined randomization scheme kept only in the pharmacy. The study will be blinded to ordering and treating providers, as well as the RA and nurse. The investigators will use an online randomization tool, and randomization will be even between the two groups. S An ED nurse will place an IV catheter if the patient does not already have one, and will record heart rate, blood pressure, respiratory rate, oxygen saturation immediately before the infusion and 5 minutes after. The medication will be given over 2 minutes by a nurse, who will remain in the room for 5 minutes after infusion. The patient will remain on pulse oximeter for 30 minutes. The RA or study investigator will administer a post-infusion survey to document any adverse effects and will record pre- and post-infusion vital signs 5 minutes after infusion. The IV catheter will then be removed unless required for another clinical indication as determined by the treating physician. After the 30 minute monitoring period, the patient will resume standard ED care and can be transferred to the psychiatric ED or CAPS whenever the bed is available. The RA or investigator will administer follow up depression and SI scales after 1 hour, 3 hours, 1 day, 3 days, and 7 days either in the psychiatric ED or CAPS, or by telephone if the patient has been discharged.

ELIGIBILITY:
Inclusion Criteria:

* Determined, based upon medical and social work evaluation, to require inpatient psychiatric admission without further need for medical diagnostic evaluation and treatment.
* Treatment-resistant depression (defined as failure of response to trials of at least 2 antidepressant courses, each of at least 4 weeks' duration)
* Parent/guardian available for consent (in person or by phone)

Exclusion Criteria:

* Any of the following co-existing diagnoses: primary psychotic disorder (schizophrenia, schizoaffective) autism spectrum disorder, developmental delay/intellectual disability, substance abuse disorder within the last 6 months
* Aggressive behavior, homicidal ideation
* Altered mental status
* Pregnancy or breastfeeding,
* Currently receiving (or receipt within last 24 hours) medication acting on NMDA receptor system (lamotrigine, dextromethorphan, methadone, clarithromycin, amantadine)
* Incomplete medical evaluation or stabilization
* Contraindications to or anaphylaxis or prior adverse reaction to Ketamine
* No caregiver available
* In custody of a law enforcement agency

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Beck Depression Inventory Depression sub-scale Score | 1 hour, 3 hours, 1 day, 3 days, 7 days after treatment
  Beck depression inventory score, 0-20 (higher score associated with worse depression)

SECONDARY OUTCOMES:
Change in Beck Depression Inventory anxiety sub-scale score | 1 hour, 3 hours, 1 day, 3 days, 7 days after treatment
  Depression sub-score, 0-20 (higher score associated with worse anxiety)
Change in Beck Depression Inventory self-concept sub-scale score | 1 hour, 3 hours, 1 day, 3 days, 7 days after treatment
  Depression sub-score, 0-20 (higher score associated with worse self-concept)
Change in Suicidal Ideation Questionnaire score | 1 hour, 3 hours, 1 day, 3 days, 7 days after treatment
  Suicidal Ideation score, 0-120 (higher score associated with higher suicide risk)

CONTACTS AND LOCATIONS:
Locations (1):
- Rady Children's Hospital San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
Study data will be published in the future